CLINICAL TRIAL: NCT05187143
Title: Clinical and Radiographic Outcomes of a New Fully Tapered Implant With the One-time One-abutment Approach: In-line Clinical Case Series With 1-year Follow-up
Brief Title: Results of a New Fully Tapered Implant at One Year
Status: Completed | Type: Observational
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Juan Blanco Carrión, 1. Periodontology Unit, School of Medicine and Dentistry, University of Santiago de Compostela, Spain., University of Santiago de Compostela
Other Study IDs: SC_BLX_US19
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Implant Site Reaction
Keywords: Fully tapered implants, platform switching, one-time one-abutment, crestal bone loss.
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: DENTAL IMPLANT — The study implants were 3.5, 3.75 or 4.5 mm implant diameter, Straumann® BLX implant SLActive® Roxolid® (Institut Straumann AG, Basel, Switzerland) and the abutment was a 0 °, 2.5 mm of height Straumann® Screw-retained Abutment. The length of the implants was 6, 8 and 10 mm. The 6 mm implant is only commercially available in 3.75 and 4.5 diameter.

SUMMARY:
Objective: The aim of this prospective observational clinical study is to evaluate the bone level changes in a new implant design, fully tapered and platform switching with the one-time one-abutment protocol after one year of loading.

Material and methods: Thirty patients received 1 or 2 implants (6, 8 and 10 mm in length, 3.5, 3.75 or 4.5 mm diameter and bone level design) to replace a single or multiple gap. Radiographic, clinical, esthetic and survival success rate were evaluated after one year of loading.

Results: At 12 months post final loading, there were no peri-implant bone loss in any of the cases. Mean marginal crestal bone loss between surgery and crown placement was 0.19 ± 0.17 (p <0.0001). Between surgery and 12 months of follow-up, the mean marginal crestal bone loss was 0.25 ± 0.24 (p <0.0001). There were a SSD between 1 year follow-up and crown placement in PI in the mesial (0.33 ± 0.54 p= 0.003) and distal aspect (0.5 ± 0.73 p= 0.001). The PPD was SSD deeper at 1 year follow-up than at crown placement only in the mesial and distal probing (averaged depth=0.75 and p<0.0005). No statistically significant differences were found for any of the other clinical and est

ELIGIBILITY:
Inclusion Criteria:

* Males or females with, at least 18 years old.
* Single and multiple gaps (premolars & molars) that require single and partial fixed restorations (2 implants, 1 pontic).
* Adequate bone quantity at the implant site to allow the placement of diameter 3.5, 3.75 or 4.5 mm and lengths of 6 mm, 8 mm, 10 mm, 12 mm or 14 mm.
* Patients had to be informed of the follow up visits and willing to attend to the clinical centre for these appointments.

Exclusion Criteria:

As systemic exclusion criteria, patients with systemic diseases that could interfere with dental implant therapy, smokers of more than 10 cigarettes per day, alcoholism or drug abuse, physical or mental disabilities, pregnant or lactating women and/or conditions or circumstances, in the opinion of the investigator, that could prevent the completion of the participation in the study or interfering with the analysis of study results (non-compliance).

The presence of one of the following circumstances was considered a local exclusion criterion: patients with inadequate oral hygiene (plaque control > 25%) (Mombelli et al., 1987), untreated endodontic lesions, any bone augmentation procedure before or during the implant placement, local inflammation (including untreated periodontitis), mucosal diseases such as erosive lichen planus, history of local irradiation therapy in the head-neck area and/or extraction sockets with less than 12 weeks of healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 30 patients (30 implants) were included (19 male and 11 female). All patients completed the follow-up at one year.
  All patients had periodontal health. Implants were placed in 22 non-smoking patients and 8 light smokers. At the time of surgery, there were no complications in any patient.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Bone level changes | One year
  To assess changes in interproximal bone levels, standardized periapical radiographs were taken of the treated areas.

CONTACTS AND LOCATIONS:
Locations (1):
- Master Periodoncia, Santiago de Compostela, Spain

IPD SHARING:
Plan to Share IPD: No